CLINICAL TRIAL: NCT05645705
Title: Two-Week Clinical Safety and Saliva Flow Quantification
Brief Title: A Two-Week Study of Clinical Safety and Saliva Flow Quantification
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johnson & Johnson Consumer Inc. (J&JCI) (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CCSORC005121; CCSORC005121 (Other: Johnson & Johnson Consumer Inc. (J&JCI))
Record Dates: First submitted 2022-12-01; First posted 2022-12-09 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-09

CONDITIONS: Healthy
MeSH Terms: interventions — Ethanol

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Arm 1: Brush/ LISTERINE Cool Mint Antiseptic Mouthwash (Experimental): At Day 0, participants will use their products at the site and saliva samples will be taken at pre-determined timepoints. At home, participants will use their products twice a day for approximately 14 days.
  Interventions: Other: Colgate Cavity Protection Toothpaste; Other: LISTERINE Cool Mint Antiseptic Mouthwash
- Arm 2: Brush / Listerine Advanced Gum Alcohol (Experimental): At Day 0, participants will use their products at the site and saliva samples will be taken at pre-determined timepoints. At home, participants will use their products twice a day for approximately 14 days.
  Interventions: Other: Colgate Cavity Protection Toothpaste; Other: Listerine Advanced Gum Alcohol
- Arm 3: Brush / Listerine Advanced Gum Zero (Experimental): At Day 0, participants will use their products at the site and saliva samples will be taken at pre-determined timepoints. At home, participants will use their products twice a day for approximately 14 days.
  Interventions: Other: Colgate Cavity Protection Toothpaste; Other: Listerine Advanced Gum Zero
- Arm 4: Brush / LISTERINE ULTRACLEAN Tartar Control Antiseptic Mouthwash Cool Mint (Experimental): At Day 0, participants will use their products at the site and saliva samples will be taken at pre-determined timepoints. At home, participants will use their products twice a day for approximately 14 days.
  Interventions: Other: Colgate Cavity Protection Toothpaste; Other: LISTERINE ULTRACLEAN Tartar Control Antiseptic Mouthwash Cool Mint
- Arm 5: Brush Only (Other): At Day 0, participants will use their products at the site and saliva samples will be taken at pre-determined timepoints. At home, participants will use their products twice a day for approximately 14 days.
  Interventions: Other: Colgate Cavity Protection Toothpaste

INTERVENTIONS:
Other: Colgate Cavity Protection Toothpaste — Participants will use Colgate Cavity Protection Toothpaste for brushing teeth twice daily.
Other: LISTERINE Cool Mint Antiseptic Mouthwash — Participants will use 20 mL of LISTERINE Cool Mint Antiseptic Mouthwash for 30 seconds after brushing twice daily.
  Arms: Arm 1: Brush/ LISTERINE Cool Mint Antiseptic Mouthwash
Other: Listerine Advanced Gum Alcohol — Participants will use 20 mL of Listerine Advanced Gum Alcohol Rinse for 30 seconds after brushing twice daily.
  Arms: Arm 2: Brush / Listerine Advanced Gum Alcohol
Other: Listerine Advanced Gum Zero — Participants will use 20 mL of Listerine Advanced Gum Zero Rinse for 30 seconds after brushing twice daily.
  Arms: Arm 3: Brush / Listerine Advanced Gum Zero
Other: LISTERINE ULTRACLEAN Tartar Control Antiseptic Mouthwash Cool Mint — Participants will use 20 mL of LISTERINE ULTRACLEAN Tartar Control Antiseptic Mouthwash Cool Mint Rinse for 30 seconds after brushing twice daily.
  Arms: Arm 4: Brush / LISTERINE ULTRACLEAN Tartar Control Antiseptic Mouthwash Cool Mint

SUMMARY:
The purpose of this study is to assess the oral tissue tolerance (tissues within the mouth) for irritation caused by added ingredients in mouthwashes. This will be assessed based on oral tissue exams and adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

* Able to comprehend and follow the requirements and restrictions of the study (including willingness to use the assigned study products per instructions, availability on scheduled visit dates and likeliness of completing the clinical study) based upon research site personnel's assessment
* Evidence of a personally signed and dated informed consent document indicating the participant (or legally acceptable representative) has been informed of all pertinent aspects of the trial
* Able to read and understand the local language (participant is capable of reading the documents)
* Adequate oral hygiene (that is, brush teeth daily and exhibit no signs of oral neglect)
* Adults, 18 years of age and older, in good general and oral health without any known allergy to commercial dental products or cosmetics
* Evidence of being fully vaccinated for corona virus disease-2019 (COVID-19) (adults 60 years and older)
* Negative pregnancy urine tests (females of child-bearing potential only)
* Females of childbearing potential must be using a medically acceptable method of birth control for at least one month prior to Visit 1 and agree to continue using this method during their participation in the study
* Resting baseline unstimulated salivary sample must be equal to or greater than 0.3 milliliter per minute (mL/min) to continue in the study
* A minimum of 20 natural teeth with scorable facial and lingual surfaces. Teeth that are grossly carious, extensively restored, orthodontically banded, abutments, exhibiting severe generalized cervical and/or enamel abrasion, or third molars will not be included in the tooth count
* Absence of significant oral soft tissue pathology, excluding plaque-induced gingivitis, based on a visual examination and at the discretion of the Investigator
* Absence of advanced periodontitis based on a clinical examination and discretion of the dental examiner
* Absence of fixed or removable orthodontic appliance or removable partial dentures

Exclusion Criteria:

* History of significant adverse effects, including sensitivities or suspected allergies, following use of oral hygiene products such as toothpastes, mouthwashes and red food dye
* Dental prophylaxis within four weeks prior to Baseline visit
* History of medical conditions requiring prophylactic antibiotic coverage prior to invasive dental procedures
* Use of antibiotics, anti-inflammatory or anticoagulant therapy, phenytoin sodium or diphenylhydantoin, cyclosporin A, immunostimulants/ immunomodulators during the study or within the one month prior to the Baseline exam. Intermittent use of certain anti-inflammatory medication (ibuprofen, Aspirin); oral steroids and calcium channel blockers are acceptable at the discretion of the investigator
* Use of chemotherapeutic anti-plaque/anti-gingivitis products such as triclosan, essential oils, cetylpyridinium chloride, sodium fluoride with CPC, stannous fluoride, zinc or chlorhexidine digluconate containing mouthwashes and toothpastes within the four weeks prior to the Baseline exam
* Known allergy or sensitivity or history of significant adverse effects to any of the investigational product and/or product ingredients (or other ingredients in the products)
* Self-reported pregnancy or lactation (this criterion is due to oral tissue changes related to pregnancy and nursing which can affect interpretation of study results)
* Self-reported smokeless tobacco user including snuff, chewing tobacco, vaping and e-cigarette usage
* Males with a pregnant partner or a partner who is currently trying to become pregnant
* Suspected alcohol or substance abuse (examples, amphetamines, benzodiazepines, cocaine, marijuana, opiates)
* Significant medical or oral condition which may interfere with a participant's participation in the study, including cancer, chronic kidney disease, chronic obstructive pulmonary disease (COPD), immunocompromised state (weakened immune system) from solid organ transplant, serious heart conditions, (such as heart failure, coronary artery disease, or cardiomyopathies) Sickle cell disease, Type 2 diabetes mellitus at the discretion of the Investigator
* Participation in any clinical trial within 30 days of Screening visit
* Diagnosed Temporo-mandibular joint dysfunction/disorder
* Participants who wear bruxing devices, dental aligners, retainers
* Participants who were previously screened and ineligible or were randomized to receive investigational product
* Participants who are related to those persons involved directly or indirectly with the conduct of this study (that is, principal investigator, sub-investigators, study coordinators, other site personnel, employees of Johnson & Johnson subsidiaries, contractors of Johnson & Johnson, and the families of each)
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the participant inappropriate for entry into this study
* COVID-19 restrictions: participants who fail to meet the criteria of the site's screening consent for Preventing Infection in the site's COVID-19 consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2022-11-28 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Oral Tolerance Based on Oral Hard and Soft Tissue Exams | Baseline up to Day 14
  Change from baseline in oral tolerance based on oral had and soft tissue exams will be reported. Oral examination will be conducted to monitor oral soft and hard tissues tolerance to the treatments. Buccal and sublingual mucosae, lips/labial mucosa, mucobuccal fold, gingiva, tongue, hard and soft palate, uvula, oropharynx, teeth and dental restorations will be examined and findings will be recorded in the electronic data capture (EDC) system.
Number of Participants with Adverse Events (AEs) | Up to Day 14
  An AE is any untoward medical occurrence in a clinical study participant temporally associated with the clinical investigation, whether or not the event has a causal relationship to the participant's participation in the trial.

SECONDARY OUTCOMES:
Salivary Flow Rate | Baseline and immediately (0), 2, 5, 10, 15 and 30 minutes after intervention use
  Saliva samples will be collected by participants at baseline and then immediately (0), 2, 5, 10, 15 and 30 minute timepoints after intervention. The final amount of saliva will be weighed to calculate the milliliter per minute (mL/min). The saliva flow rate will be expressed as mL/min.
Saliva Potential of Hydrogen (pH) | Baseline and 2, 5, 10, 15 and 30 minutes after intervention use
  The pH value of saliva will be measured by placing the saliva sample onto the pH-sensitive electrode.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery Milleman, DDS, Principal Investigator — Salus Research, Inc.
Locations (1):
- Salus Research, Inc., Fort Wayne, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Consumer Inc. has an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu

REFERENCES:
- [Derived] Milleman K, Bosma ML, Saito A, Gorecki P, Ding Y, DelSasso A, Wills K, Milleman JL. Comparison of safety, salivary flow rate, and pH with different mouthrinse formulations in addition to toothbrushing vs toothbrushing only: Results from a 2-week phase 4 randomized controlled clinical trial. J Am Dent Assoc. 2025 Dec;156(12):991-1000.e3. doi: 10.1016/j.adaj.2025.08.022. PMID 41338687
- See also: Two-Week Clinical Safety and Saliva Flow Quantification — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CCSORC005121&attachmentIdentifier=31680829-5987-4328-87b9-5c1be8e6ab4d&fileName=CCSORC005121_CSR_Synopsis.pdf&versionIdentifier=